CLINICAL TRIAL: NCT06939530
Title: Comparision of Hydrodilatation Results at Different Volumes in Adhesive Capsulitis by Phases.
Acronym: HYCAFVOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Muñoz Paz (Other)
Collaborators: Universidad de Córdoba (Other); Maimonides Institute for Biomedical Research of Cordoba (IMIBIC) (Unknown); Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Sponsor-Investigator, Javier Muñoz Paz, Medical intern resident in physical medicine and rehabilitation, Maimónides Biomedical Research Institute of Córdoba
Organization: Maimónides Biomedical Research Institute of Córdoba (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HYCAFVOL
Record Dates: First submitted 2025-04-01; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Capsulitis of Shoulder; Hydrodilatation
Keywords: Adhesive Capsulitis; frozen shoulder; hydrodilatation; suprascapular nerve block
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Ensayo clínico aleatorizado por bloques en paralelo con triple cegamiento.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For this trial, we propose triple blinding. The principal investigator, Javier Muñoz, will be the only one aware of the treatment assignment. Neither the patient, the reviewer, the physiotherapists, nor the statistician will be aware of the treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adhesive Capsulitis Phase 1 (Active Comparator): Adhesive Capsulitis Phase 1 --> Patients in phase 1 will be considered as those in which the predominant clinical picture is pain accompanied by limitation of ROM
  Interventions: Procedure: Hydrodilatation (20 ml); Procedure: Hydrodilatation (40 ml)
- Adhesive Capsulitis Phase 2 (Active Comparator): Adhesive Capsulitis Phase 2 --> Patients in whom ROM limitation predominates in the face of pain.
  Interventions: Procedure: Hydrodilatation (20 ml); Procedure: Hydrodilatation (40 ml)

INTERVENTIONS:
Procedure: Hydrodilatation (20 ml) — First, an SSNB will be performed with 4 ml of 0.25% anesthetic + 0.5 ml of corticosteroid in the suprascapular notch.
  After 15 minutes of the SSNB, ultrasound-guided HD will begin. To do this, the patient will be placed in a lateral decubitus position on the unaffected arm. The arm to be treated will be positioned at the patient's side without forcing its extension. The joint cavity will then be approached posteriorly, introducing a spinal needle in the ultrasound plane between the humeral cortex and the labrum. The joint cavity will then be confirmed by introducing physiological saline solution and observing its reflux by pushing the plunger. Subsequently, 5 ml of 0.25% anesthetic + 0.5 ml of corticosteroid will be introduced, and the corresponding volume will be completed with saline solution, this case 20 ml.
Procedure: Hydrodilatation (40 ml) — First, an SSNB will be performed with 4 ml of 0.25% anesthetic + 0.5 ml of corticosteroid in the suprascapular notch.
  After 15 minutes of the SSNB, ultrasound-guided HD will begin. To do this, the patient will be placed in a lateral decubitus position on the unaffected arm. The arm to be treated will be positioned at the patient's side without forcing its extension. The joint cavity will then be approached posteriorly, introducing a spinal needle in the ultrasound plane between the humeral cortex and the labrum. The joint cavity will then be confirmed by introducing physiological saline solution and observing its reflux by pushing the plunger. Subsequently, 5 ml of 0.25% anesthetic + 0.5 ml of corticosteroid will be introduced, and the corresponding volume will be completed with saline solution, this case 40 ml.

SUMMARY:
Adhesive capsulitis (AC) causes a global limitation of active and passive range of motion (ROM) in the shoulder, with or without pain, and no other radiographic findings. The natural process is self-limiting, evolving in three or four phases. It is common in women around 50 years of age. Diagnosis is based on clinical symptoms, with imaging tests being nonspecific. Treatment options include physical therapy (PT), intra-articular corticosteroid injections, suprascapular nerve block (SSNB), and hydrodilatation (HD). The latter is useful for expanding and reducing inflammation of the joint capsule through insufflation with saline solution, anesthetics, and corticosteroids.

Objectives: To determine whether patients with AC, stratified by phase, who receive high-volume HD therapy achieve better outcomes in the Shoulder Pain and Disability Index (SPADI), Analgesic Analogue Scale (VAS), and ROM at the first, third, and sixth months of therapy compared to patients who receive low-volume HD. To determine whether there are differences in FST times and to determine mean axilar recess (AR) values.

Methods: A randomized, triple-blind, parallel-block clinical trial will be conducted in 64 patients with AC in phases 1 and 2, aged 30 to 70 years, with limited active and passive ROM in two planes, and shoulder pain lasting more than 3 months. HD will be administered with volumes of 20 ml or 40 ml, followed by a physical therapy program. Outcomes will be reviewed at the first, third, and sixth months of HD. Variables collected will include SPADI, VAS, ROM, Lattinen assessment, AR size, and time to completion of PT

ELIGIBILITY:
Inclusion Criteria:

* Ages between 30 and 70 years.
* Limited ROM, both active and passive, in two planes.
* Shoulder pain lasting more than 3 months.

Exclusion Criteria:

* Lidocaine + trial with improved ROM.
* Conditions that preclude treatment (active cancer, tissue infection, oral anticoagulant use, cardiac arrhythmias, etc.)
* Previously receiving HD treatment in less than 1 year.
* Stage 0 or 3 AC.
* Non-adherence to the PT program, with attendance failures exceeding 20%.
* Presence of conditions that can cause similar symptoms, such as acromioclavicular osteoarthritis, labral injury, massive rotator cuff tear, or rheumatic diseases.
* Intra-articular corticosteroid injection in less than 2 months.
* Technique failure.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder pain and disability index (SPADI) | Initial and 1 - 3 - 6 month after hydrodilatation
  The Shoulder Pain Disability Index is a widely used outcome measure in studies that provides information about pain and limitation of shoulder pathologies.
  * Pain Scale How severe is the pain? 0 = no pain and 10 = the worst pain imaginable.
    * At its worst?
    * When lying on that side?
    * When reaching for something on a high shelf?
    * When touching the back of your neck?
    * When pushing with the affected arm?
  * Disability Scale:
  How much difficulty do you have? 0 = no pain and 10 = the worst pain imaginable.
  * Washing your hair.
  * Washing your back.
  * Putting on a T-shirt or sweater.
  * Putting on a button-down shirt.
  * Putting on your pants.
  * Placing an object on a high shelf.
  * Lifting a heavy object weighing 4.5 kilograms.
  * Taking something from his back pocket.
  Then, pain and disability are obtained separately, and a percentage of impairment is combined.
  This index has demonstrated "good internal consistency, convergent validity, and reliability" in its Spanish version.
Visual Analgesic Scale (VAS) | Initial and 1 - 3 - 6 month after hydrodilatation
  The VAS "is a validated subjective measure for acute and chronic pain." It allows for the measurement of pain intensity with maximum reproducibility.
  It consists of a 10-centimeter horizontal line, with the extreme expressions of a symptom at each end. To the left (0) is the absence or lowest intensity, and to the right (10) is the highest intensity. The patient is asked to mark the point on the line that indicates the intensity. The minimally detectable differences for the symptom level to be acceptable are 2 to 3 points.
Range of motion assessment (ROM) | Initial and 1 - 3 - 6 month after hydrodilatation
  Range of motion assessment is a basic practice in the study of shoulder pathologies, especially in the case of AC. ROM should be measured, both actively and passively.
  The ROMs that will be assessed actively and passively will primarily be flexion, abduction, external rotation (with the arm at 90° of abduction, by asking the patient to show us the palm of their hand), and internal rotation (with the arm at 90° of abduction, by asking the patient to show us the back of their hand). All of these are measured with the PLURIMETER inclinometer.

SECONDARY OUTCOMES:
Axillary recess (AR) size | Initial
  This will be measured using ultrasound with a longitudinal section of the AR. The patient will be placed supine with the shoulder abducted at 90° and the elbow flexed.
Time from star to end of physiotherapy | From 1 session to a maximum of 3 months of PT
  They will begin the PT program in less than 3-5 days. The PT start and start date will be scheduled according to pre-established criteria.
  The following criteria will be established for discontinuing PT treatment:
  * No improvement of 15% in ROM after full HD after 16 sessions.
  * Recovery of full ROM after 4 sessions.
  * Increased pain that makes PT impossible.
  * Maximum of 24 PT sessions.
  It will be measured in days.

OTHER OUTCOMES:
Lattinen Test | Initial and 1 - 3 - 6 month after hydrodilatation
  The Lattinen test is a widely used tool for assessing pain, validated in Spain as a tool to measure the degree of pain in patients with chronic pain. This scale consists of five items scored from 0 to 4:
  1. Pain intensity.
  2. Pain frequency.
  3. Analgesic use.
  4. Degree of disability.
  5. Hours of sleep.
  Although this test is widely used in chronic pain conditions, its use in AC is not very common. However, we believe it can provide important data such as analgesic medication intake. This is why we consider its use appropriate.
Patient Global Patient Improvement Impression Scale (PGI-I) | It will be measured at the last check-up 6 months after HD
  The PGI-I consists of a single question that asks the patient to classify the relief obtained with the treatment according to a 7-point Likert scale: "much better"; "much better"; "a little better"; "no change"; "a little worse"; "much worse"; "much worse".
Global CGI - GI Impression of Global Improvement Scale (CGI - GI) | It will be measured at the last check-up 6 months after HD
  The CGI-I, the physician compares the patient's initial clinical condition with the current condition: "Compared to the patient's condition at the time of admission to the project [prior to the start of medication], this patient's condition is: 1=much better since the start of treatment; 2=much improved; 3=minimally improved; 4=no change since baseline (the start of treatment); 5=minimally worse; 6=much worse; 7=much worse since the start of treatment."

CONTACTS AND LOCATIONS:
Overall Officials: Javier Muñoz Paz, degree in medicine, Principal Investigator — Hospital Universitario Reina Sofia de Cordoba; Fernando J Mayordomo Riera, Head of service, Study Director — Hospital Universitario Reina Sofia de Cordoba; Jose Peña Amaro, Professor of Histology - UCO, Study Director — Universidad de Córdoba
Locations (1):
- Hospital Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stella SM, Gualtierotti R, Ciampi B, Trentanni C, Sconfienza LM, Del Chiaro A, Pacini P, Miccoli M, Galletti S. Ultrasound Features of Adhesive Capsulitis. Rheumatol Ther. 2022 Apr;9(2):481-495. doi: 10.1007/s40744-021-00413-w. Epub 2021 Dec 23. PMID 34940958
- [Background] González-Escalada JR, Camba A, Muriel C, Rodríguez M, Contreras D, De Barutell C. Validación del índice de Lattinen para la evaluación del paciente con dolor crónico. Vol. 19, Rev Soc Esp Dolor. 2012.
- [Background] Vicente Herrero MT, Delgado Bueno S, Bandrés Moyá F, Ramírez Iñiguez de la Torre MV, Capdevila García L. Valoración del dolor. Revisión Comparativa de Escalas y Cuestionarios. Revista de la Sociedad Española del Dolor. 2018.
- [Background] Membrilla-Mesa MD, Cuesta-Vargas AI, Pozuelo-Calvo R, Tejero-Fernandez V, Martin-Martin L, Arroyo-Morales M. Shoulder pain and disability index: cross cultural validation and evaluation of psychometric properties of the Spanish version. Health Qual Life Outcomes. 2015 Dec 21;13:200. doi: 10.1186/s12955-015-0397-z. PMID 26690943
- [Background] Paruthikunnan SM, Shastry PN, Kadavigere R, Pandey V, Karegowda LH. Intra-articular steroid for adhesive capsulitis: does hydrodilatation give any additional benefit? A randomized control trial. Skeletal Radiol. 2020 May;49(5):795-803. doi: 10.1007/s00256-019-03316-8. Epub 2019 Dec 17. PMID 31844950
- [Background] Lin CL, Lee YH, Chen YW, Liao CD, Huang SW. Predictive Factors of Intra-articular Corticosteroid Injections With Ultrasound-Guided Posterior Capsule Approach for Patients With Primary Adhesive Capsulitis. Am J Phys Med Rehabil. 2024 Mar 1;103(3):215-221. doi: 10.1097/PHM.0000000000002340. Epub 2023 Sep 22. PMID 37752075
- [Background] Lee JH, Lee JH, Chang MC. Association of Range of Motion Deficit and Recurrence of Pain After Treatment of Adhesive Capsulitis. Pain Ther. 2024 Apr;13(2):241-249. doi: 10.1007/s40122-024-00578-6. Epub 2024 Feb 5. PMID 38315379
- [Background] de Sire A, Agostini F, Bernetti A, Mangone M, Ruggiero M, Dinatale S, Chiappetta A, Paoloni M, Ammendolia A, Paolucci T. Non-Surgical and Rehabilitative Interventions in Patients with Frozen Shoulder: Umbrella Review of Systematic Reviews. J Pain Res. 2022 Aug 19;15:2449-2464. doi: 10.2147/JPR.S371513. eCollection 2022. PMID 36016536
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Shanahan EM, Gill TK, Briggs E, Hill CL, Bain G, Morris T. Suprascapular nerve block for the treatment of adhesive capsulitis: a randomised double-blind placebo-controlled trial. RMD Open. 2022 Nov;8(2):e002648. doi: 10.1136/rmdopen-2022-002648. PMID 36418088
- [Background] Jung TW, Lee SY, Min SK, Lee SM, Yoo JC. Does Combining a Suprascapular Nerve Block With an Intra-articular Corticosteroid Injection Have an Additive Effect in the Treatment of Adhesive Capsulitis? A Comparison of Functional Outcomes After Short-term and Minimum 1-Year Follow-up. Orthop J Sports Med. 2019 Jul 23;7(7):2325967119859277. doi: 10.1177/2325967119859277. eCollection 2019 Jul. PMID 31384617
- [Background] Pimenta M, Vassalou EE, Klontzas ME, Dimitri-Pinheiro S, Ramos I, Karantanas AH. Ultrasound-guided hydrodilatation for adhesive capsulitis: capsule-preserving versus capsule-rupturing technique. Skeletal Radiol. 2024 Feb;53(2):253-261. doi: 10.1007/s00256-023-04392-7. Epub 2023 Jul 3. PMID 37400605
- [Background] Whelan G, Yeowell G, Littlewood C. Patient experiences of hydrodistension as a treatment for frozen shoulder: A longitudinal qualitative study. PLoS One. 2024 Jun 14;19(6):e0304236. doi: 10.1371/journal.pone.0304236. eCollection 2024. PMID 38875237
- [Background] Swaroop S, Gupta P, Patnaik S, Reddy SS. Intra-articular Steroid alone vs Hydrodilatation with intra-articular Steroid in Frozen Shoulder - A Randomised Control Trial. Malays Orthop J. 2023 Mar;17(1):34-39. doi: 10.5704/MOJ.2303.005. PMID 37064640
- [Background] Vita F, Pederiva D, Tedeschi R, Spinnato P, Origlio F, Faldini C, Miceli M, Stella SM, Galletti S, Cavallo M, Pilla F, Donati D. Adhesive capsulitis: the importance of early diagnosis and treatment. J Ultrasound. 2024 Sep;27(3):579-587. doi: 10.1007/s40477-024-00891-y. Epub 2024 Jun 6. PMID 38844748
- [Background] Cho JH. Updates on the treatment of adhesive capsulitis with hydraulic distension. Yeungnam Univ J Med. 2021 Jan;38(1):19-26. doi: 10.12701/yujm.2020.00535. Epub 2020 Aug 31. PMID 32862630
- [Background] Dimitri-Pinheiro S, Klontzas ME, Vassalou EE, Pimenta M, Soares R, Karantanas AH. Long-Term Outcomes of Ultrasound-Guided Hydrodistension for Adhesive Capsulitis: A Prospective Observational Study. Tomography. 2023 Oct 14;9(5):1857-1867. doi: 10.3390/tomography9050147. PMID 37888739
- [Background] Poku D, Hassan R, Migliorini F, Maffulli N. Efficacy of hydrodilatation in frozen shoulder: a systematic review and meta-analysis. Br Med Bull. 2023 Sep 12;147(1):121-147. doi: 10.1093/bmb/ldad018. PMID 37496207
- [Background] Rex SS, Kottam L, McDaid C, Brealey S, Dias J, Hewitt CE, Keding A, Lamb SE, Wright K, Rangan A. Effectiveness of interventions for the management of primary frozen shoulder : a systematic review of randomized trials. Bone Jt Open. 2021 Sep;2(9):773-784. doi: 10.1302/2633-1462.29.BJO-2021-0060.R1. PMID 34555926
- [Background] Buchbinder R, Green S, Youd JM, Johnston RV, Cumpston M. Arthrographic distension for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD007005. doi: 10.1002/14651858.CD007005. PMID 18254123
- [Background] Wang JC, Tsai PY, Hsu PC, Huang JR, Wang KA, Chou CL, Chang KV. Ultrasound-Guided Hydrodilatation With Triamcinolone Acetonide for Adhesive Capsulitis: A Randomized Controlled Trial Comparing the Posterior Glenohumeral Recess and the Rotator Cuff Interval Approaches. Front Pharmacol. 2021 May 7;12:686139. doi: 10.3389/fphar.2021.686139. eCollection 2021. PMID 34025441
- [Background] Makki D, Al-Yaseen M, Almari F, Monga P, Funk L, Basu S, Walton M. Shoulder hydrodilatation for primary, post-traumatic and post-operative adhesive capsulitis. Shoulder Elbow. 2021 Oct;13(6):649-655. doi: 10.1177/1758573220977179. Epub 2020 Dec 9. PMID 34804214
- [Background] Fares MY, Koa J, Abboud JA. Assessment of therapeutic clinical trials for adhesive capsulitis of the shoulder. JSES Int. 2023 Jan 31;7(3):412-419. doi: 10.1016/j.jseint.2023.01.003. eCollection 2023 May. PMID 37266176
- [Background] Patel R, Urits I, Wolf J, Murthy A, Cornett EM, Jones MR, Ngo AL, Manchikanti L, Kaye AD, Viswanath O. A Comprehensive Update of Adhesive Capsulitis and Minimally Invasive Treatment Options. Psychopharmacol Bull. 2020 Oct 15;50(4 Suppl 1):91-107. doi: 10.64719/pb.4384. PMID 33633420
- [Background] Hill JL. Evidence for Combining Conservative Treatments for Adhesive Capsulitis. Ochsner J. 2024 Spring;24(1):47-52. doi: 10.31486/toj.23.0128. PMID 38510216
- [Background] Do JG, Hwang JT, Yoon KJ, Lee YT. Correlation of Ultrasound Findings With Clinical Stages and Impairment in Adhesive Capsulitis of the Shoulder. Orthop J Sports Med. 2021 May 10;9(5):23259671211003675. doi: 10.1177/23259671211003675. eCollection 2021 May. PMID 33997079
- [Background] Lee BC, Yeo SM, Do JG, Hwang JH. Sequential Ultrasound Assessment of Peri-Articular Soft Tissue in Adhesive Capsulitis of the Shoulder: Correlations with Clinical Impairments-Sequential Ultrasound in Adhesive Capsulitis. Diagnostics (Basel). 2022 Sep 15;12(9):2231. doi: 10.3390/diagnostics12092231. PMID 36140631
- [Background] Dimitriou D, Winkler E, Zindel C, Grubhofer F, Wieser K, Bouaicha S. Is routine magnetic resonance imaging necessary in patients with clinically diagnosed frozen shoulder? Utility of magnetic resonance imaging in frozen shoulder. JSES Int. 2022 Jun 11;6(5):855-858. doi: 10.1016/j.jseint.2022.05.009. eCollection 2022 Sep. PMID 36081696
- [Background] Erber B, Hesse N, Goller S, Gilbert F, Ricke J, Glaser C, Heuck A. Diagnostic performance and interreader agreement of individual and combined non-enhanced and contrast-enhanced MR imaging parameters in adhesive capsulitis of the shoulder. Skeletal Radiol. 2024 Feb;53(2):263-273. doi: 10.1007/s00256-023-04391-8. Epub 2023 Jul 3. PMID 37400604
- [Background] Ammerman BM, Dennis ER, Ling D, Hannafin JA. Ultrasound-Guided Glenohumeral Corticosteroid Injection for the Treatment of Adhesive Capsulitis of the Shoulder: The Role of Clinical Stage in Response to Treatment. Sports Health. 2024 May-Jun;16(3):333-339. doi: 10.1177/19417381231168799. Epub 2023 Apr 25. PMID 37097090
- [Background] Schiltz M, Goudman L, Moens M, Nijs J, Hatem SM. The diagnostic value of physical examination tests in adhesive capsulitis: a systematic review. Eur J Phys Rehabil Med. 2023 Dec;59(6):724-730. doi: 10.23736/S1973-9087.23.07940-6. Epub 2023 Sep 22. PMID 37737049
- [Background] Picasso R, Pistoia F, Zaottini F, Marcenaro G, Miguel-Perez M, Tagliafico AS, Martinoli C. Adhesive Capsulitis of the Shoulder: Current Concepts on the Diagnostic Work-Up and Evidence-Based Protocol for Radiological Evaluation. Diagnostics (Basel). 2023 Nov 9;13(22):3410. doi: 10.3390/diagnostics13223410. PMID 37998547
- [Background] Dimitri-Pinheiro S, Pinto BS, Pimenta M, Neves JS, Carvalho D. Influence of diabetes on response to ultrasound guided hydrodistension treatment of adhesive capsulitis: a retrospective study. BMC Endocr Disord. 2022 Sep 12;22(1):227. doi: 10.1186/s12902-022-01144-x. PMID 36096804
- [Background] Chuang SH, Chen YP, Huang SW, Kuo YJ. Association between adhesive capsulitis and thyroid disease: a meta-analysis. J Shoulder Elbow Surg. 2023 Jun;32(6):1314-1322. doi: 10.1016/j.jse.2023.01.033. Epub 2023 Mar 4. PMID 36871608
- [Background] Dyer BP, Rathod-Mistry T, Burton C, van der Windt D, Bucknall M. Diabetes as a risk factor for the onset of frozen shoulder: a systematic review and meta-analysis. BMJ Open. 2023 Jan 4;13(1):e062377. doi: 10.1136/bmjopen-2022-062377. PMID 36599641
- [Background] Abudula X, Maimaiti P, Yasheng A, Shu J, Tuerxun A, Abudujilili H, Yang R. Factors associated with frozen shoulder in adults: a retrospective study. BMC Musculoskelet Disord. 2024 Jun 26;25(1):493. doi: 10.1186/s12891-024-07614-8. PMID 38926699
- [Background] Fields BKK, Skalski MR, Patel DB, White EA, Tomasian A, Gross JS, Matcuk GR Jr. Adhesive capsulitis: review of imaging findings, pathophysiology, clinical presentation, and treatment options. Skeletal Radiol. 2019 Aug;48(8):1171-1184. doi: 10.1007/s00256-018-3139-6. Epub 2019 Jan 3. PMID 30607455
- [Background] Date A, Rahman L. Frozen shoulder: overview of clinical presentation and review of the current evidence base for management strategies. Future Sci OA. 2020 Oct 30;6(10):FSO647. doi: 10.2144/fsoa-2020-0145. PMID 33312703
- [Background] Mezian K, Coffey R, Chang KV. Frozen Shoulder(Archived). 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482162/ PMID 29489251
- [Background] Mertens MG, Meeus M, Verborgt O, Girbes EL, Horno SM, Aguilar-Rodriguez M, Duenas L, Navarro-Ledesma S, Fernandez-Sanchez M, Luque-Suarez A, Struyf F. Exploration of the clinical course of frozen shoulder: A longitudinal multicenter prospective study of functional impairments. Braz J Phys Ther. 2023 Jul-Aug;27(4):100539. doi: 10.1016/j.bjpt.2023.100539. Epub 2023 Aug 23. PMID 37639942
- [Background] Li D, St Angelo JM, Taqi M. Adhesive Capsulitis (Frozen Shoulder). 2025 Mar 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532955/ PMID 30422550
- See also: Frozen shoulder adhesive capsulitis - UpToDate — https://www.uptodate.com/contents/frozen-shoulder-adhesive-capsulitis?search=Hudnall%20S.%20Frozen%20shoulder%20%28adhesive%20capsulitis%29.%202024.%20UpToDate.%20&source=search_result&selectedTitle=1%7E150&usage_type=default&display_rank=1
- See also: Physical examination of the shoulder- UpToDate — https://www.uptodate.com/contents/physical-examination-of-the-shoulder?search=Stephen%20S%2C%20Dixon%20B.%20Physical%20examination%20of%20the%20shoulder.%202024.%20&source=search_result&selectedTitle=1%7E150&usage_type=default&display_rank=1

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT06939530/Prot_SAP_000.pdf
  • Informed Consent Form: INFORMED CONSENT AND PATIENT INFORMATION SHEET (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT06939530/ICF_001.pdf